CLINICAL TRIAL: NCT06098469
Title: Developping a a Brain-controlled Art App to Ease Residual Symptoms of Depression
Acronym: DEEPBLUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: API/2019/102
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neurofeedback (Experimental): 10 neurofeedback sessions + depressive rating scales
  Interventions: Device: Neurofeedback sessions

INTERVENTIONS:
Device: Neurofeedback sessions — 10 Neurofeedback sessions, psychiatric interview (MADRS, QIDS-C16), reverse-correlation task, QIDS-SR16, EQ-5D-5L, motivation assessment

SUMMARY:
The study evaluate the effect of 10 neurofeedback sessions on the residual symptoms of depressive patients in partial remission.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 25 to 65 included
* Information and signed informed consent
* Patients with a diagnosis of major depressive episode in remission
* MADRS score between 14 and 22
* Patients with residual symptoms as assessed by MADRS items
* No cognitive impairment.
* Right-handed

Exclusion Criteria:

* Subjects with legal incapacity or limited legal capacity
* Subjects unlikely to cooperate with the study and/or poor cooperation anticipated by the investigator
* Pregnant women
* Subjects in the exclusion period of another study or is on the "national volunteer list".
* Subjects with another psychiatric pathology (bipolar mood disorder, psychosis, obsessive-compulsive disorder, addictive pathology, schizophrenia)
* Subjects under a protective measure such as guardianship or safeguard of justice.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of 10 neurofeedback sessions on residual symptoms in depressive patients in partial remission | Week 10
  Reduction in MADRS score to < 8 (complete remission) after 10 neurofeedback sessions, in particular cumulative score less than or equal to 2 for hedonic and fatigue dimensions

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel HAFFEN, MD PhD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU Besançon, Besançon, France